CLINICAL TRIAL: NCT05934409
Title: Improved Adipose Tissue Storage of Dietary Fatty Acids as a New Mechanism for the Rapid Remission of Hepatic and Cardiac Metabolic Dysfunction After Bariatric Surgery
Brief Title: Adipose Tissue Storage in the Rapid Remission of Hepatic and Cardiac Metabolic Dysfunction After Bariatric Surgery
Acronym: CB5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Carpentier, Tenure professor, Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-4624
Record Dates: First submitted 2023-06-08; First posted 2023-07-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Bariatric surgery; remission from Type 2 diabetes; PET imaging; adipose tissue
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bariatric Surgery; Niacin

STUDY DESIGN:
Intervention Model Description: It will be a randomized crossover study prior to bariatric surgery (visits A0 and A1) followed by a longitudinal follow-up study after surgery (visits B0 and C0) in two groups (type 2 diabetes vs. controls). Inside each group, the protocol will be carried out as a within-subject, in which each subject will serve as his/her own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): without T2D according to Diabetes Canada diagnostics criteria:
  Interventions: Procedure: Bariatric surgery; Drug: Nicotinic Acid
- group with Type 2 diabetes (Experimental): with T2D according to Diabetes Canada diagnostics criteria:
  Interventions: Procedure: Bariatric surgery; Drug: Nicotinic Acid

INTERVENTIONS:
Procedure: Bariatric surgery — Laparoscopic Sleeve Gastrectomy
Drug: Nicotinic Acid — Only during A1. 150mg every half hour for 6 hours. A total dose of 1800mg will be ingested.
  Other Names: Niacin

SUMMARY:
The present protocol aims to understand and establish whether there is a causal link between adipose tissue metabolic remodeling and Type 2 Diabetes (T2D) remission after bariatric surgery.

All participants will have a bariatric surgery, divided in 2 groups: with or without T2D.

DETAILED DESCRIPTION:
This clinical assay will include 5 visits: the screening visit and four 9-hour postprandial metabolic sessions (A0, A1, B0 and C0) before and after surgery:

* initial visit: screening
* before surgery: 2 metabolic sessions A0 and A1 (without/with niacin) will be performed, in random order, at least one week interval.
* 12 days post surgery: 1 metabolic session B0 (without niacin)
* 1 year post surgery: 1 metabolic session C0 (without niacin)

Each metabolic visit will last 9 hours with:

* perfusion of stable tracers,
* ingestion of a liquid meal
* Positron-Emitting-Tomography (PET) acquisitions using radiopharmaceuticals such as [18F]-fluoro-6-thia-heptadecanoic acid ([18F]-FTHA) and [11C]-palmitate,
* MRI acquisitions.[18F]fluoro-6-thia-heptadecanoic acid (FTHA).

The niacin will be given during metabolic visits A1 as a regulator of lipids metabolism. During these visits, the subjects will ingest 150mg every half hour for 6 hours. Niacin will be used as a pharmacological suppressor of dietary fatty acid (DFA) spillover in order to determine the role played by this mechanism in the reduction of postprandial endogen glucose production (EGP) in T2D after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65
* BMI 35 kg/m2
* Diagnosed T2D - according to Diabetes Canada diagnostics criteria.
* Diagnosed non-T2D - according to Diabetes Canada diagnostics criteria.
* Women with a negative serum pregnancy test.

Exclusion Criteria:

* Treatment with an oral contraceptive;
* Treatment with fibrate, thiazolidinedione, insulin, or beta-blocker, drugs that affect metabolism and cannot be stopped temporarily or which have long-lasting effects;
* Presence of overt cardiovascular disease, liver or renal failure or other uncontrolled medical conditions;
* Any other contraindication to surgery or to temporarily suspending current medications for diabetes, lipids or hypertension;
* Smoking or consumption of more than 2 alcoholic beverages per day;
* Any contraindication to MRI;
* A Diabetes Remission (DiaRem) score >8 (low probability of T2D remission);
* Having participated to a research study with exposure to radiation in the last two years before the start of the study;
* Pregnant or breastfeeding women;
* Patients weighing more than 200 kg to respect the weight and gantry limit of our MRI and PET/CT scanners.
* Being allergic to eggs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in white adipose tissue dietary fatty acid (DFA) trapping and partitioning | measured after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  [18F]-FTHA PET
Change in lean organ (liver, heart and muscle) DFA uptake and partitioning | measured after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  [18F]-FTHA PET
Change in liver non-esterified fatty acid (NEFA) uptake, oxidation, esterification and secretion into very low-density lipoprotein (VLDL). | measured before and after liquid meal at Baseline (A0), at Day 12 (B0) and at Week 52 (C0)
  calculated from the same multicompartmental equation using liver [11C]-palmitate kinetics
Change in Endogenous Glucose production and meal glucose systemic flux | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  i.v. and oral stable isotope tracer
Change in cardiac non-esterified fatty acid (NEFA) uptake, oxidation and esterification | measured before and after liquid meal at Baseline (A0), at Day 12 (B0) and at Week 52 (C0)
  calculated from the same multicompartmental equation using cardiac [11C]-palmitate kinetics

SECONDARY OUTCOMES:
Change in plasma NEFA flux | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  calculated from i.v. stable isotope tracer (mass spectrometry).
Change in hepatic Triglyceride (TG) content | measured at Baseline (A0), at Day 12 (B0) and at Week 52 (C0)
  magnetic resonance imaging (MRI)
Change in insulin secretion | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  Determined by measuring C-peptide kinetics following the liquid meal
Change in total substrate utilisation | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  measured by using indirect calorimetry
Change in gene and protein expression of white adipose tissue (WAT) | measured at Baseline (A0), at Day 12 (B0) and at Week 52 (C0)
  WAT biopsy
Change in hormonal response | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  Multiplex assay
Change in insulin resistance /sensitivity | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  Determined by measuring circulating glucose, NEFA and insulin following the liquid meal
Change in histology of white adipose tissue (WAT) | measured at Baseline (A0), at Day 12 (B0) and at Week 52 (C0)
  WAT biopsy
Change in metabolite response | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0
  Colorimetric assay
Change in plasma distribution of DFA metabolites (WAT DFA spillover) | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  calculated from i.v. and oral stable isotope tracers (mass spectrometry) incorporated into triglyceride-rich lipoproteins and NEFA.
Change in glycerol turnover | measured before and after liquid meal at Baseline (A0 +A1), at Day 12 (B0) and at Week 52 (C0)
  calculated from [1,1,2,3,3-2H]-glycerol i.v.

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- centre de recherche du CHUS, Sherbrooke, Quebec, Canada